CLINICAL TRIAL: NCT07081594
Title: Investigating the Impact of Sex Hormones on Corticospinal Excitability, Motor Learning, and Fatigue in Females With Multiple Sclerosis
Brief Title: Investigating the Impact of Sex Hormones in Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Milap Sandhu (Other)
Responsible Party: Sponsor-Investigator, Milap Sandhu, Principle Investigator, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Other Study IDs: STU00224323
Record Dates: First submitted 2025-06-17; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Sex hormones; menstrual cycle
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-Menopausal Women: Naturally cycling women with multiple sclerosis

SUMMARY:
Emerging evidence indicates that females with MS experience worsened symptoms during the luteal phase (post ovulation) of the menstrual cycle when progesterone levels rise and estradiol fluctuate. The rapid hormonal swings may disrupt hypothalamic regulation, leading to an increase in body temperature - a well-established trigger for MS symptom exacerbation. These hormonal changes could also affect neuromuscular function, as estradiol and progesterone receptors are present in the nervous system and skeletal muscles.

Three critical aspects of motor rehabilitation are corticospinal excitability, motor learning, and fatigability. Previous research indicates that corticospinal excitability and the capacity to learn fine motor tasks fluctuate across menstrual cycles, indicating hormonal influences on neuroplasticity. However, it remains unclear how these hormonal fluctuations specifically affect corticospinal excitability, motor learning, and motor fatigability in females with MS. Understanding these relationships could significantly improve rehabilitation approaches. For example, pre-menopause females with MS may experience a more optimal state for neuroplasticity during the follicular phase of their cycles, therefore providing a potential window for greater rehabilitation efficacy.

DETAILED DESCRIPTION:
The objective of this project is to systematically examine how hormonal fluctuations pre-menopause influence corticospinal excitability, motor learning, and motor fatigability in females with MS. The study is structured around the following specific aims:

Aim 1: Quantify the effects of estradiol and progesterone levels on corticospinal excitability in pre- menopausal females with MS. We will elicit motor evoked potentials by cortical and subcortical stimulation of corticospinal axons using transcranial magnetic stimulation (TMS).

Aim 2: Evaluate how hormonal fluctuations across menstrual phases impact motor learning ability in pre-menopause females with MS. Participants will be asked to perform a finger sequence motor learning task using visual feedback. The task will be performed using a computer keyboard. Participants will be asked to copy the numerical sequence on a monitor in front of them that pertains to a number on the keyboard with their fingers. Participants will be given three different sequences with equivalent difficulty at each session to avoid carry-over effects between visits.

Aim 3: Determine the relationship between hormonal fluctuations and motor fatigability in pre-menopause females with MS. Participants will perform a maximal voluntary force (MVF). Participants will then be asked to pinch to 80% of their MVF, and maintain this hold for as long as possible1. The trial will end when the force drops below 40% MVF. Two trials in total will be performed. Average time to fatigue (40% MVF) and slope of the drop-off will be calculated as a measure of overall fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of relapsing-remitting, primary progressive or secondary progressive MS with no minimum years since diagnosis
* Stable disease modifying therapies for at least 6 months
* Eumenorrheic females

Exclusion Criteria:

* Another diagnosis (e.g., peripheral neuropathies or orthopedic)
* Pregnancy as confirmed by urine test
* Irregular menstrual cycles
* Diagnosis of premenstrual dysphoric disorder or polycystic ovary syndrome
* Taking antipsychotic medications / does not pass the TMS safety checklist

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with menstrual cycles and any form of multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Corticospinal excitability | At 3 points during the individual's 1-month menstrual cycle, 1) Early Follicular 2) Late Follicular 3) Luteal
  Measuring the brain to muscle connection using transcranial magnetic stimulation - a non-invasive way to measure brain activity. Peak to Peak amplitude in mV is recorded
Blood Draw | At 3 points during the individual's 1-month menstrual cycle, 1) Early Follicular 2) Late Follicular 3) Luteal
  To quantify estradiol and progesterone levels. Normative values of estradiol (E) and progesterone (P) per phase: early follicular (E: 125pmol/L; P: 0.38nmol/L), late follicular (E: 464pmol/L; P: 0.188nmol/L), luteal (E: 412pmol/L; P: 28.8nmol/L)

SECONDARY OUTCOMES:
strength | At 3 points during the individual's 1-month menstrual cycle, 1) Early Follicular 2) Late Follicular 3) Luteal
  Measured by a pinch maximal voluntary contraction in lb-f
Fatigue | At 3 points during the individual's 1-month menstrual cycle, 1) Early Follicular 2) Late Follicular 3) Luteal
  Measured with a pinch fatiguing task to estimate how quickly muscle of the hand fatigues. Measured in Seconds
Motor Learning | At 3 points during the individual's 1-month menstrual cycle, 1) Early Follicular 2) Late Follicular 3) Luteal
  A visuomotor tracking task to measure difference between target trace and performed trace, measured in root mean squared error

CONTACTS AND LOCATIONS:
Overall Officials: Milap Sandhu, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be available after completion of the study upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following IRB approval, documents will be available
Access Criteria: These data will be available upon request

REFERENCES:
- [Background] Christogianni A, O'Garro J, Bibb R, Filtness A, Filingeri D. Heat and cold sensitivity in multiple sclerosis: A patient-centred perspective on triggers, symptoms, and thermal resilience practices. Mult Scler Relat Disord. 2022 Nov;67:104075. doi: 10.1016/j.msard.2022.104075. Epub 2022 Jul 25. PMID 35963205
- [Background] Karim HT, Huppert TJ, Erickson KI, Wollam ME, Sparto PJ, Sejdic E, VanSwearingen JM. Motor sequence learning-induced neural efficiency in functional brain connectivity. Behav Brain Res. 2017 Feb 15;319:87-95. doi: 10.1016/j.bbr.2016.11.021. Epub 2016 Nov 11. PMID 27845228
- [Background] Casamento-Moran A, Mooney RA, Chib VS, Celnik PA. Cerebellar Excitability Regulates Physical Fatigue Perception. J Neurosci. 2023 Apr 26;43(17):3094-3106. doi: 10.1523/JNEUROSCI.1406-22.2023. Epub 2023 Mar 13. PMID 36914263
- [Background] Hackney AC, ed. Sex Hormones, Exercise and Women: Scientific and Clinical Aspects. 1st ed. 2017. Springer International Publishing : Imprint: Springer; 2017. doi:10.1007/978-3-319-44558-81
- [Background] Gilli F, DiSano KD, Pachner AR. SeXX Matters in Multiple Sclerosis. Front Neurol. 2020 Jul 3;11:616. doi: 10.3389/fneur.2020.00616. eCollection 2020. PMID 32719651